CLINICAL TRIAL: NCT03289182
Title: Post-Marketing Surveillance of MabThera Subcutaneous in Patients With Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: An Observational Study of MabThera Subcutaneous (SC) Safety in Participants With Non-Hodgkin's Lymphoma (NHL) or Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39600
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MabThera: Participants with NHL will be administered 1400 milligrams (mg) and those with with CLL will be administered 1600 mg MabThera subcutaneously at the discretion of the physician in accordance with local clinical practice and local labeling, and will be observed for 6 years.
  Interventions: Drug: MabThera

INTERVENTIONS:
Drug: MabThera — Participants will be administered MabThera 1400 mg (NHL) or 1600 mg (CLL) at the discretion of the physician in accordance with local clinical practice and local labeling.

SUMMARY:
This is a prospective, multicenter, non-interventional study to test the safety and effectiveness of MabThera administered subcutaneously in participants with NHL or CLL. The length of study is expected to be 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants administered with MabThera subcutaneously within the approved indication in Korea
* Participants previously untreated with MabThera subcutaneously

Inclusion Criteria for NHL participants for MabThera subcutaneously 1400mg:

* Relapsed or chemoresistant follicular lymphoma (FL) (B, C, and D type by international working formulation classification of B-cell NHL) participants
* Previously untreated FL participants in combination with chemotherapy
* Participants who are treated with maintenance therapy after the treatment of FL participants responding to induction therapy.
* Cluster of differentiation 20-positive, diffuse large B-cell NHL participants in combination with cyclophosphamide, doxorubicin, vincristine, and prednisolone (8 cycles) chemotherapy

Inclusion Criteria for CLL participants for MabThera subcutaneously 1600mg:

- Previously untreated or relapsed/refractory CLL participants in combination with chemotherapy

Exclusion Criteria:

* Pregnant or breastfeeding women
* Participants who are out of locally approved indications, dosage, and administration including medication error
* Contraindication in use by locally approved indications, dosage, and administration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving treatment for NHL or CLL with MabThera SC under observation according to standard of care and in line with the current local labelling in Korea.
Sampling Method: Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline up to Year 6

SECONDARY OUTCOMES:
Percentage of Participants with Overall Response as Assessed by the Investigator Using the Cheson 2014 Criteria for NHL | Baseline up to Year 6
Percentage of Participants with Overall Response as Assessed by the Investigator Using the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 Criteria | Baseline up to Year 6

CONTACTS AND LOCATIONS:
Locations (25):
- South Korea (25):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center; Hematology, Daegu
  - Chungnam National University Hospital, Daejeon
  - Korea University Ansan Hospital, Gyeonggi-do
  - St. Vincent's Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital; Department of Hematology, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Inje University, Sanggye-Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Seoul National University Hospital; Department of Oncology, Seoul
  - Severance Hospital, Yonsei University Health System; Oncology, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
  - St. Mary'S Hospital, the Catholic University School of Medicine; Internal Medicine, Seoul
  - Korea Cancer Center Hospital; Surgery, Seoul
  - Korea University Guro Hospital; Department of Hematology & Oncology, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan